CLINICAL TRIAL: NCT01949766
Title: Transition From Buphenyl to RAVICTI for the Therapy of Byler Disease
Status: No longer available | Type: Expanded Access
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO12070385.2
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Byler Disease
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1 | interventions — glycerol phenylbutyrate

INTERVENTIONS:
Drug: Glycerol phenylbutyrate
  Other Names: RAVICTI

SUMMARY:
This is a single patient compassionate use protocol to determine whether RAVICTI will improve bile flow in a subject who previously tolerated therapy with Buphenyl.

ELIGIBILITY:
Inclusion Criteria:

* Byler Disease
* Cholestasis
* Tolerance of Buphenyl therapy

Exclusion Criteria:

* Allergy/Hypersensitivity to RAVICTI

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult